CLINICAL TRIAL: NCT02404493
Title: A Clinical Trial to Evaluate the Efficacy of an Investigational Nighttime Moisturizing Balm in the Management of Mild to Moderate Atopic Dermatitis in Infants and Toddlers
Brief Title: Test to Determine the Effectiveness of Moisturizing Balm Used on Babies With Dry, Itchy Skin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of subject enrollment and the eczema season has completed
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CO-141020101115-THCT
Record Dates: First submitted 2015-03-18; First posted 2015-03-31 (Estimated); Results first posted 2017-03-24 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-02

CONDITIONS: Eczema
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Eczema; Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EpiCeram Skin Barrier Emulsion (Active Comparator): Marketed. Apply in a thin layer to the affected skin areas two times per day (or as needed) and massage gently into the skin.
  Interventions: Device: EpiCeram Skin Barrier Emulsion
- 1% Colloidal Oatmeal Balm (Experimental): Not Yet Marketed. Apply in a thin layer to the affected skin areas at least once at night or more if needed (anytime), and massage gently into the skin.
  Interventions: Drug: 1% Colloidal Oatmeal Balm

INTERVENTIONS:
Device: EpiCeram Skin Barrier Emulsion — EpiCeram Skin Barrier Emulsion
  Arms: EpiCeram Skin Barrier Emulsion
Drug: 1% Colloidal Oatmeal Balm — Experimental Product 1% Colloidal Oatmeal Balm
  Other Names: Eczema Moisturizing Balm
  Arms: 1% Colloidal Oatmeal Balm

SUMMARY:
The purpose of this 3 week study is to test the effectiveness of an over-the-counter (OTC) skin balm in infants and toddlers with mild to moderate dry, itchy skin.

DETAILED DESCRIPTION:
50 infants and toddlers will be enrolled in this study to yield 40 completed subjects, 30 babies in the active treatment group and 10 babies in the positive control group.

Infants and toddlers aged 6 to 47 months inclusive will receive either a prescription or non-marketed investigational product for the treatment of eczema. Caregivers will be asked to stop use of prescription eczema treatments one week before the start of the study and during the study. Caregivers will apply study product to babies as indicated for 14 days to affected areas.

Subject caregivers will record treatment use in a daily diary and complete questionnaires. A dermatologist will examine and score the babies eczema and symptoms. Skin moisture levels will also be tested.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and follow the requirements of the study (including availability on scheduled visit dates)
2. Male or female of any race or ethnicity, 6 months to 47 months of age;
3. Diagnosed as having eczema
4. Willing to stop use of all non-assigned moisturizers and/or creams for the entire duration of the study
5. Child must have bedtime/sleep issues due to their dry, itchy skin

Exclusion Criteria:

1. Use of a therapeutic (over-the-counter or prescription) body wash that contains an active ingredient for eczema
2. Participation in any clinical study within 30 days of Visit 1
3. Active infection of any type at the start of the study
4. Diagnosed as having severe eczema
5. Atopic Dermatitis requiring systemic, super-potent (Class I) or potent (Class II or III) topical corticosteroids
6. Child wakes up 3 or more times during the night
7. Child is awake more than 60 minutes during the night
8. Child sleeps for less than a total of 9 hours (during the day or night)
9. Child requires greater than 2.0 mg per day of inhaled or intranasal corticosteroids

Ages: 6 Months to 47 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amisha Parikh-Das, PhD, Study Director — Johnson & Johnson Consumer Inc. (J&JCI); Ethlynn Schorr, MD, Principal Investigator — TKL Research, Inc.
Locations (1):
- TKL Research, Fair Lawn, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1% Colloidal Oatmeal Balm: 1% colloidal oatmeal balm applied in a thin layer to affected skin areas at least once at night or more if needed
- EpiCeram Skin Barrier Emulsion: EpiCeram skin barrier emulsion applied in a thin layer to affected skin areas two times per day or as needed
Period: Overall Study
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Started | 17 | 6
Completed | 16 | 5
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion | Total
Number analyzed (Participants) | 17 | 6 | 23
Age, Continuous [Mean (Standard Deviation); unit: months] | 21.8 (9.66) | 22.5 (10.78) | 22.0 (9.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 0 | 7
  Male | 10 | 6 | 16
Region of Enrollment [Number; unit: participants]
  USA | 17 | 6 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Corneometer Measurement Immediately Following Treatment
Description: Corneometer is a non-invasive instrument that measures hydration on the skin surface. During assessment, the corneometer was placed at a site adjacent to affected skin areas. Corneometer readings are directly related to the skin's electrical capacitance and increase as the skin becomes more hydrated.
Time Frame: Day 0 - Pretreatment (Baseline) to Day 0 - immediately post treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
arbitrary units | 656.31 (273.322) | 234.72 (176.566)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; The null hypothesis was no difference between the baseline score and the post-baseline score. The alternative hypothesis was a difference between the baseline score and the post-baseline score; Test type: Superiority or Other; p < 0.001, One-sample t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.023, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.003, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 422.81, 95% CI 2-sided [166.435 to 679.186], Standard Error of Mean 122.905

2. Primary Outcome: Change From Baseline in Mean Corneometer Measurement 12 Hours After Treatment
Description: as for outcome 1
Time Frame: Day 0 - Pretreatment (Baseline) to 12 Hours After treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
arbitrary units | 55.12 (47.124) | 2.11 (15.629)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.754, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.013, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Median Difference (Final Values) = 52.30, 95% CI 2-sided [12.230 to 92.373], Standard Error of Mean 19.210

3. Secondary Outcome: Change From Baseline in Mean Corneometer Measurement 24 Hours After Treatment
Description: as for outcome 1
Time Frame: Day 0 - Pretreatment (Baseline) to 24 Hours After treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
arbitrary units | 178.35 (138.651) | 14.83 (29.347)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.271, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.002, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 167.95, 95% CI 2-sided [67.046 to 268.854], Standard Error of Mean 48.210

4. Secondary Outcome: Change From Baseline in Mean Corneometer Measurement 3 Days After Treatment
Description: as for outcome 1
Time Frame: Day 0 - Pretreatment (Baseline) to 3 Days After treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
arbitrary units | 226.85 (244.028) | 8.17 (15.769)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.002, One-sample t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.260, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.040, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 221.97, 95% CI 2-sided [11.254 to 432.680], Standard Error of Mean 100.674

5. Secondary Outcome: Change From Baseline in Mean Corneometer Measurement 7 Days After Treatment
Description: as for outcome 1
Time Frame: Day 0 - Pretreatment (Baseline) to 7 Days After treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
arbitrary units | 208.52 (169.098) | 17.50 (30.615)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.220, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.011, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 194.00, 95% CI 2-sided [50.712 to 337.291], Standard Error of Mean 68.461

6. Secondary Outcome: Change From Baseline in Mean Corneometer Measurement 14 Days After Treatment
Description: as for outcome 1
Time Frame: Day 0 - Pretreatment (Baseline) to 14 Days After treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
arbitrary units | 158.65 (170.627) | 23.60 (20.298)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.002, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.060, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.107, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 134.90, 95% CI 2-sided [-32.266 to 302.063], Standard Error of Mean 79.567

7. Secondary Outcome: Eczema Area and Severity Index (EASI) on Day 1 - Change From Baseline
Description: The surface and severity of eczema is measured using the Eczema Area and Severity Index (EASI). A regional body surface area tabulation based on severity ranging from 0 (absent) to 3 (severe), and severity of signs of disease, then multiplied by body area with final calculation ranging from 0-72.
Time Frame: Day 0 - Pretreatment (Baseline) to Day 1
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
units on a scale | 0.04 (0.434) | -0.12 (0.436)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.692, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.541, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.492, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.250 to 0.502], Standard Error of Mean 0.180

8. Secondary Outcome: Eczema Area and Severity Index (EASI) on Day 3 - Change From Baseline
Description: as for outcome 7
Time Frame: Day 0 - Pretreatment (Baseline) to Day 3
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
units on a scale | -0.54 (0.802) | -0.48 (0.852)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.017, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.223, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.518, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.635 to 0.331], Standard Error of Mean 0.231

9. Secondary Outcome: Eczema Area and Severity Index (EASI) on Day 7 - Change From Baseline
Description: as for outcome 7
Time Frame: Day 0 - Pretreatment (Baseline) to Day 7
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
units on a scale | -0.73 (0.884) | -0.15 (1.544)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.005, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.821, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.060, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-1.435 to 0.032], Standard Error of Mean 0.351

10. Secondary Outcome: Eczema Area and Severity Index (EASI) on Day 14 - Change From Baseline
Description: as for outcome 7
Time Frame: Day 0 - Pretreatment (Baseline) to Day 14
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
units on a scale | -0.74 (0.962) | -0.85 (0.814)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.007, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.051, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.926, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.410 to 0.375], Standard Error of Mean 0.188

11. Secondary Outcome: Investigator's Global Atopic Dermatitis Assessment (IGADA) on Day 1 - Change From Baseline
Description: The signs and symptoms of eczema are measured using the Investigator's Global Atopic Dermatitis Assessment (IGADA). An assessment of atopic dermatitis based on a 4 point scale, ranging from 0 (absent) to 3 (severe), is used to describe signs and symptoms in 4 designated body regions. Based on the presence or absence of the total number of signs and symptoms, the final rating is categorized as clear, almost clear, mild, moderate, severe, or very severe.
Time Frame: Day 0 - Pretreatment (Baseline) to Day 1
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
units on a scale | -0.1 (0.44) | -0.2 (0.41)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.580, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.363, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.539, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.531 to 0.286], Standard Error of Mean 0.20

12. Secondary Outcome: Investigator's Global Atopic Dermatitis Assessment (IGADA) on Day 3 - Change From Baseline
Description: as for outcome 11
Time Frame: Day 0 - Pretreatment (Baseline) to Day 3
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
units on a scale | -0.3 (0.60) | -0.5 (0.55)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.055, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.076, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.682, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.672 to 0.449], Standard Error of Mean 0.27

13. Secondary Outcome: Investigator's Global Atopic Dermatitis Assessment (IGADA) on Day 7 - Change From Baseline
Description: as for outcome 11
Time Frame: Day 0 - Pretreatment (Baseline) to Day 7
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
units on a scale | -0.4 (0.51) | -0.7 (0.52)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.004, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.025, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.991, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.509 to 0.514], Standard Error of Mean 0.24

14. Secondary Outcome: Investigator's Global Atopic Dermatitis Assessment (IGADA) on Day 14 - Change From Baseline
Description: as for outcome 11
Time Frame: Day 0 - Pretreatment (Baseline) to Day 14
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
units on a scale | -0.6 (0.51) | -1.0 (0.00)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.334, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.214 to 0.600], Standard Error of Mean 0.19

15. Secondary Outcome: Dryness Scale Score on Day 1 - Change From Baseline
Description: An assessment of dryness based on a 4 point scale, ranging from 0 (none) to 4 (severe dryness).
Time Frame: Day 0 - Pretreatment (Baseline) to Day 1
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 9 | 4
units on a scale | -0.2 (0.44) | 0.0 (0.00)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.169, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.317, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.778 to 0.278], Standard Error of Mean 0.24

16. Secondary Outcome: Dryness Scale Score on Day 3 - Change From Baseline
Description: An assessment of dryness based on a 4 point scale, ranging from 0 (none) to 4 (severe dryness).
Time Frame: Day 0 - Pretreatment (Baseline) to Day 3
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 9 | 4
units on a scale | -0.9 (0.33) | -0.5 (0.58)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.182, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.027, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.931 to -0.069], Standard Error of Mean 0.19

17. Secondary Outcome: Dryness Scale Score on Day 7 - Change From Baseline
Description: An assessment of dryness based on a 4 point scale, ranging from 0 (none) to 4 (severe dryness).
Time Frame: Day 0 - Pretreatment (Baseline) to Day 7
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 9 | 4
units on a scale | -1.2 (0.44) | -1.3 (0.96)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.080, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.699, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.824 to 0.574], Standard Error of Mean 0.31

18. Secondary Outcome: Dryness Scale Score on Day 14 - Change From Baseline
Description: An assessment of dryness based on a 4 point scale, ranging from 0 (none) to 4 (severe dryness).
Time Frame: Day 0 - Pretreatment (Baseline) to Day 14
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 9 | 4
units on a scale | -1.2 (0.44) | -1.5 (1.00)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.058, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.711, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.607 to 0.857], Standard Error of Mean 0.33

19. Secondary Outcome: Caregiver's Itch Assessment on Day 3 - Change From Baseline
Description: An assessment of dryness based on the following scale, 0 (don't have an opinion), 1 (none), 2 (a little), 3 (a lot), 4 (all the time).
Time Frame: Day 0 - Pretreatment (Baseline) to Day 3
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 15 | 6
units on a scale | -0.73 (0.884) | -1.00 (0.632)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.006, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.012, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.932, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.391 to 0.424], Standard Error of Mean 0.194

20. Secondary Outcome: Caregiver's Itch Assessment on Day 7 - Change From Baseline
Description: as for outcome 19
Time Frame: Day 0 - Pretreatment (Baseline) to Day 7
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 15 | 6
units on a scale | -0.87 (0.915) | -1.17 (0.408)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.003, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.767, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.410 to 0.547], Standard Error of Mean 0.228

21. Secondary Outcome: Caregiver's Itch Assessment on Day 14 - Change From Baseline
Description: as for outcome 19
Time Frame: Day 0 - Pretreatment (Baseline) to Day 14
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 15 | 5
units on a scale | -1.00 (0.845) | -1.20 (0.447)
Statistical Analysis 1: Comparison: 1% Colloidal Oatmeal Balm; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 2: Comparison: EpiCeram Skin Barrier Emulsion; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.004, One sample t-test — The significance level threshold level was 0.05
Statistical Analysis 3: Comparison: 1% Colloidal Oatmeal Balm vs EpiCeram Skin Barrier Emulsion; The null hypothesis was no difference between groups. The alternative hypothesis was a difference between groups; Test type: Superiority or Other; p = 0.571, ANCOVA — The significance level threshold level was 0.05; Change from baseline as response, baseline score as covariate and treatment as factor; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.650 to 0.370], Standard Error of Mean 0.242

22. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 0 Pretreatment (Baseline) - Responder Role
Description: Questions were answered before treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: What is the role of the responder?
Time Frame: 0 Days Pretreatment (Baseline)
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  Father | 0 | 0
  Mother | 100 | 100
  Grandparent | 0 | 0
  Other | 0 | 0

23. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 0 Pretreatment (Baseline) - Sleeping Arrangement
Description: Questions were answered before treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: What is the sleeping arrangement?
Time Frame: 0 Days Pretreatment (Baseline)
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  Infant crib separate room | 23.5 | 33.3
  Infant crib parent's room | 41.2 | 0
  In parent's bed | 17.6 | 50.0
  Infant crib in room with sibling | 0 | 0
  Other | 17.6 | 16.7

24. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 0 Pretreatment (Baseline) - Time Child Usually Put to Bed
Description: Questions were answered before treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: What time do you usually put your child to bed at night? Time is represented as post meridiem (pm).
Time Frame: 0 Days Pretreatment (Baseline)
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: hours.minutes
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
hours.minutes | 9.04 (1.16) | 9.10 (0.35)

25. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 0 Pretreatment (Baseline) - Difficulty of Bedtime
Description: Questions were answered before treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: Typically, how difficult is bedtime for your child? Caregiver answered based on a 5 point system ranging from 'very easy' to 'very difficult'.
Time Frame: 0 Days Pretreatment (Baseline)
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  Very easy | 5.9 | 16.7
  Somewhat easy | 52.9 | 50.0
  Somewhat difficult | 17.6 | 16.7
  Moderately difficult | 17.6 | 0
  Very difficult | 5.9 | 16.7

26. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 0 Pretreatment (Baseline) - Time for Child to Fall Asleep
Description: Questions were answered before treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: How long does it typically take your child to fall asleep?
Time Frame: 0 Days Pretreatment (Baseline)
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
minutes | 27.6 (11.74) | 27.5 (15.08)

27. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 0 Pretreatment (Baseline) - Number of Times Child Awakes During the Night
Description: Questions were answered before treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: How many times does your child typically wake during the night?
Time Frame: 0 Days Pretreatment (Baseline)
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
number of times | 1.6 (1.00) | 2.3 (1.03)

28. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 0 Pretreatment (Baseline) - Total Time Child Awake During the Night
Description: Questions were answered before treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: How much total time during the night is your child typically awake?
Time Frame: 0 Days Pretreatment (Baseline)
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
minutes | 26.0 (21.85) | 44.2 (48.21)

29. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 0 Pretreatment (Baseline) - Longest Time Child is Asleep During the Night
Description: Questions were answered before treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: On average, what is the longest stretch of time that your child is asleep during the night without waking up?
Time Frame: 0 Days Pretreatment (Baseline)
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
hours | 6.28 (2.296) | 5.58 (3.105)

30. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 0 Pretreatment (Baseline) - Total Time Child is Asleep During the Night
Description: Questions were answered before treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: On average, how much total time does your child spend sleeping during the night?
Time Frame: 0 Days Pretreatment (Baseline)
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
hours | 8.46 (1.921) | 9.08 (1.908)

31. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 0 Pretreatment (Baseline) - Number of Naps Child Takes During the Day
Description: Questions were answered before treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: On a typical day, how many naps does your child take?
Time Frame: 0 Days Pretreatment (Baseline)
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: number of naps
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
number of naps | 1.2 (0.56) | 1.0 (0.89)

32. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 0 Pretreatment (Baseline) - Total Time Child Sleeps During the Day
Description: Questions were answered before treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: Typically, how much total time does your child spend sleeping during the day?
Time Frame: 0 Days Pretreatment (Baseline)
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
hours | 2.32 (0.642) | 1.57 (1.023)

33. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 0 Pretreatment (Baseline) - Child's Sleep a Problem
Description: Questions were answered before treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: Do you consider your child's sleep a problem? Caregiver answered based on a 6 point system ranged from 'I don't have an opinion' to 'a serious problem'.
Time Frame: 0 Days Pretreatment (Baseline)
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Not a problem at all | 11.8 | 0
  A very small problem | 41.2 | 16.7
  A small problem | 23.5 | 33.3
  A moderate problem | 23.5 | 33.3
  A serious problem | 0 | 16.7

34. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 7 - Responder Role
Description: Questions were answered seven days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: What is the role of the responder?
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  Father | 0 | 0
  Mother | 100 | 100
  Grandparent | 0 | 0
  Other | 0 | 0

35. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 7- Sleeping Arrangement
Description: Questions were answered seven days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: What is the sleeping arrangement?
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  Infant crib separate room | 12.5 | 33.3
  Infant crib parent's room | 37.5 | 0
  In parent's bed | 18.8 | 50.0
  Infant crib in room with sibling | 18.8 | 0
  Other | 12.5 | 16.7

36. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 7 - Time Child Usually Put to Bed
Description: Questions were answered seven days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: What time do you usually put your child to bed at night? Time is represented as post meridiem (pm).
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: hours.minutes
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
hours.minutes | 8.46 (1.05) | 9.27 (0.40)

37. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 7 - Difficulty of Bedtime
Description: Questions were answered seven days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: Typically, how difficult is bedtime for your child? Caregiver answered based on a 5 point system ranging from 'very easy' to 'very difficult'.
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  Very easy | 6.3 | 0
  Somewhat easy | 43.8 | 50.0
  Somewhat difficult | 31.3 | 33.3
  Moderately difficult | 12.5 | 16.7
  Very difficult | 6.3 | 0

38. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 7 - Time for Child to Fall Asleep
Description: Questions were answered seven days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: How long does it typically take your child to fall asleep?
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
minutes | 28.8 (14.20) | 22.5 (12.94)

39. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 7 - Number of Times Child Awakes During the Night
Description: Questions were answered seven days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: How many times does your child typically wake during the night?
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
number of times | 1.1 (0.81) | 1.8 (1.47)

40. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 7 - Total Time Child Awake During the Night
Description: Questions were answered seven days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: How much total time during the night is your child typically awake?
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
minutes | 17.8 (11.97) | 44.2 (53.61)

41. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 7 - Longest Time Child is Asleep During the Night
Description: Questions were answered seven days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: On average, what is the longest stretch of time that your child is asleep during the night without waking up?
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
hours | 7.70 (2.206) | 6.58 (2.764)

42. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 7 - Total Time Child is Asleep During the Night
Description: Questions were answered seven days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: On average, how much total time does your child spend sleeping during the night?
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
hours | 8.81 (1.410) | 9.17 (1.633)

43. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 7 - Number of Naps Child Takes During the Day
Description: Questions were answered seven days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: On a typical day, how many naps does your child take?
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: number of naps
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
number of naps | 1.3 (0.60) | 1.2 (0.75)

44. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 7 - Total Time Child Sleeps During the Day
Description: Questions were answered seven days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: Typically, how much total time does your child spend sleeping during the day?
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
hours | 2.10 (0.649) | 2.29 (2.421)

45. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 7 - Child's Sleep a Problem
Description: Questions were answered seven days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: Do you consider your child's sleep a problem? Caregiver answered based on a 6 point system ranged from 'I don't have an opinion' to 'a serious problem'.
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Not a problem at all | 18.8 | 16.7
  A very small problem | 50.0 | 50.0
  A small problem | 18.8 | 0
  A moderate problem | 6.3 | 16.7
  A serious problem | 6.3 | 16.7

46. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 14 - Responder Role
Description: Questions were answered 14 days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: What is the role of the responder?
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
percentage of participants
  Father | 0 | 0
  Mother | 100 | 100
  Grandparent | 0 | 0
  Other | 0 | 0

47. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 14 - Sleeping Arrangement
Description: Questions were answered 14 days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: What is the sleeping arrangement?
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
percentage of participants
  Infant crib separate room | 18.8 | 20.0
  Infant crib parent's room | 37.5 | 0
  In parent's bed | 18.8 | 60.0
  Infant crib in room with sibling | 12.5 | 0
  Other | 12.5 | 20.0

48. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 14 - Time Child Usually Put to Bed
Description: Questions were answered 14 days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: What time do you usually put your child to bed at night? Time is represented as post meridiem (pm).
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: hours.minutes
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
hours.minutes | 8.48 (1.02) | 9.14 (0.31)

49. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 14 - Difficulty of Bedtime
Description: Questions were answered 14 days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: Typically, how difficult is bedtime for your child? Caregiver answered based on a 5 point system ranging from 'very easy' to 'very difficult'.
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
percentage of participants
  Very easy | 12.5 | 0
  Somewhat easy | 56.3 | 60.0
  Somewhat difficult | 25.0 | 40.0
  Moderately difficult | 6.3 | 0
  Very difficult | 0 | 0

50. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 14 - Time for Child to Fall Asleep
Description: Questions were answered 14 days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: How long does it typically take your child to fall asleep?
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
minutes | 23.8 (12.85) | 27.0 (11.51)

51. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 14 - Number of Times Child Awakes During the Night
Description: Questions were answered 14 days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: How many times does your child typically wake during the night?
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
number of times | 1.1 (0.93) | 1.6 (1.14)

52. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 14 - Total Time Child Awake During the Night
Description: Questions were answered 14 days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: How much total time during the night is your child typically awake?
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
minutes | 14.7 (9.91) | 37.0 (47.64)

53. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 14 - Longest Time Child is Asleep During the Night
Description: Questions were answered 14 days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: On average, what is the longest stretch of time that your child is asleep during the night without waking up?
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
hours | 8.19 (2.237) | 4.90 (2.966)

54. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 14 - Total Time Child is Asleep During the Night
Description: Questions were answered 14 days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: On average, how much total time does your child spend sleeping during the night?
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
hours | 8.99 (1.300) | 9.00 (2.236)

55. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 14 - Number of Naps Child Takes During the Day
Description: Questions were answered 14 days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: On a typical day, how many naps does your child take?
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: number of naps
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
number of naps | 1.2 (0.54) | 1.2 (0.84)

56. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 14 - Total Time Child Sleeps During the Day
Description: Questions were answered 14 days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: Typically, how much total time does your child spend sleeping during the day?
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
hours | 2.06 (0.722) | 1.55 (2.095)

57. Secondary Outcome: Brief Infant Sleep Questionnaire (BISQ) - Day 14 - Child's Sleep a Problem
Description: Questions were answered 14 days after treatment by the participant's caregiver. This survey collects data about sleeping venue, position, hours of sleep at night and during the day, as well as night-wakings and sleep latency. The question is: Do you consider your child's sleep a problem? Caregiver answered based on a 6 point system ranged from 'I don't have an opinion' to 'a serious problem'.
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
percentage of participants
  I don't have an opinion | 0 | 0
  Not a problem at all | 31.3 | 0
  A very small problem | 31.3 | 60.0
  A small problem | 25.0 | 20.0
  A moderate problem | 6.3 | 20.0
  A serious problem | 6.3 | 0

58. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - Skin Looks Smooth Overall
Description: Questions were answered before treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Overall, my baby's skin looks smooth".
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 29.4 | 33.3
  Somewhat disagree | 41.2 | 50.0
  Neither agree nor disagree | 11.8 | 0
  Somewhat agree | 17.6 | 0
  Strongly agree | 0 | 16.7

59. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - Skin Looks Healthy Overall
Description: Questions were answered before treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Overall, my baby's skin looks healthy".
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 5.9 | 0
  Somewhat disagree | 58.8 | 66.7
  Neither agree nor disagree | 5.9 | 0
  Somewhat agree | 23.5 | 16.7
  Strongly agree | 5.9 | 16.7

60. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - Skin Feels Soft Overall
Description: Questions were answered before treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Overall, my baby's skin feels soft".
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 23.5 | 16.7
  Somewhat disagree | 41.2 | 50.0
  Neither agree nor disagree | 17.6 | 0
  Somewhat agree | 17.6 | 0
  Strongly agree | 0 | 33.3

61. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - Baby's Skin Looks Smooth in Areas Affected by Eczema
Description: Questions were answered before treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "In the areas affected by eczema, my baby's skin looks smooth".
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 41.2 | 33.3
  Somewhat disagree | 41.2 | 50.0
  Neither agree nor disagree | 5.9 | 0
  Somewhat agree | 5.9 | 16.7
  Strongly agree | 5.9 | 0

62. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - Baby's Skin Looks Healthy in Areas Affected by Eczema
Description: Questions were answered before treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "In the areas affected by eczema, my baby's skin looks healthy".
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 11.8 | 16.7
  Somewhat disagree | 70.6 | 83.3
  Neither agree nor disagree | 0 | 0
  Somewhat agree | 11.8 | 0
  Strongly agree | 5.9 | 0

63. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - Baby's Skin Feels Soft in Areas Affected by Eczema
Description: Questions were answered before treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "In the areas affected by eczema, my baby's skin feels soft".
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 41.2 | 50.0
  Somewhat disagree | 29.4 | 33.3
  Neither agree nor disagree | 11.8 | 0
  Somewhat agree | 11.8 | 16.7
  Strongly agree | 5.9 | 0

64. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - Child's Mood Over Past Week
Description: Questions were answered before treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Over this past week, what has your child's mood been?"
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Very happy | 35.3 | 16.7
  Somewhat happy | 17.6 | 0
  No change | 17.6 | 50.0
  Somewhat fussy | 29.4 | 16.7
  Very fussy | 0 | 16.7

65. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - Child's Mood Upon Waking in Morning
Description: Questions were answered before treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Typically, how would you rate your child's mood when he/she wakes up in the morning?"
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Very happy | 23.5 | 16.7
  Somewhat happy | 35.3 | 0
  No change | 11.8 | 16.7
  Somewhat fussy | 17.6 | 50.0
  Very fussy | 11.8 | 16.7

66. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - Child Wanted to Play Over Past Week
Description: Questions were answered before treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Over this past week, how much has your child wanted to play?"
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Less than last week | 0 | 0
  No difference | 64.7 | 33.3
  A little more | 11.8 | 0
  A lot more | 0 | 16.7
  All the time | 23.5 | 50.0

67. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - Amount of Sleep Caregiver Got Over Past Week
Description: Questions were answered before treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Over this past week, how much sleep did you get at night?"
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
hours | 6.48 (1.169) | 6.19 (1.956)

68. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - Number of Times Caregiver Woke Up
Description: Questions were answered before treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "How many times did you wake up during the night?"
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
number of times | 2.2 (0.90) | 5.7 (7.06)

69. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - Amount of Time Caregiver Awake
Description: Questions were answered before treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "If you did wake up during the night, how much time were you awake (on average) before falling back asleep?"
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
hours | 0.79 (0.807) | 1.36 (0.645)

70. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - Caregiver Energy Levels Over Past Week
Description: Questions were answered before treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Over this past week, how much energy have you had to engage with your family?"
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  I don't have an opinion | 5.9 | 0
  Less than last week | 0 | 0
  No difference | 76.5 | 83.3
  A little more | 5.9 | 16.7
  A lot more | 5.9 | 0
  All the time | 5.9 | 0

71. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - How Rested Caregiver Felt Over Past Week
Description: Questions were answered before treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Over this past week, how rested have you felt?"
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  I don't have an opinion | 5.9 | 0
  Less than last week | 17.6 | 50.0
  No difference | 64.7 | 50.0
  A little more | 5.9 | 0
  A lot more | 0 | 0
  All the time | 5.9 | 0

72. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - How Alert Caregiver Felt Over Past Week
Description: Questions were answered before treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Over this past week, how alert have you felt?"
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  I don't have an opinion | 5.9 | 0
  Less than last week | 11.8 | 33.3
  No difference | 47.1 | 66.7
  A little more | 23.5 | 0
  A lot more | 0 | 0
  All the time | 11.8 | 0

73. Secondary Outcome: Caregiver Questionnaire on Day 0 Pre-treatment - How Productive Caregiver Felt Over Past Week
Description: Questions were answered before treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Over this past week, how productive have you been at work?"
Time Frame: 0 Days - Pre-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  I don't have an opinion | 23.5 | 16.7
  Less than last week | 0 | 16.7
  No difference | 64.7 | 66.7
  A little more | 5.9 | 0
  A lot more | 5.9 | 0
  All the time | 0 | 0

74. Secondary Outcome: Caregiver Questionnaire on Day 0 Post-treatment - Skin Looks Smooth Overall
Description: Questions were answered after treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Overall, my baby's skin looks smooth".
Time Frame: 0 Days - Post-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 5.9 | 0
  Somewhat disagree | 35.3 | 66.7
  Neither agree nor disagree | 17.6 | 16.7
  Somewhat agree | 23.5 | 16.7
  Strongly agree | 17.6 | 0

75. Secondary Outcome: Caregiver Questionnaire on Day 0 Post-treatment - Skin Looks Healthy Overall
Description: Questions were answered after treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Overall, my baby's skin looks healthy".
Time Frame: 0 Days - Post-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 5.9 | 0
  Somewhat disagree | 35.3 | 83.3
  Neither agree nor disagree | 11.8 | 0
  Somewhat agree | 35.3 | 16.7
  Strongly agree | 11.8 | 0

76. Secondary Outcome: Caregiver Questionnaire on Day 0 Post-treatment - Skin Feels Soft Overall
Description: Questions were answered after treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Overall, my baby's skin feels soft".
Time Frame: 0 Days - Post-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 0 | 0
  Somewhat disagree | 23.5 | 33.3
  Neither agree nor disagree | 11.8 | 33.3
  Somewhat agree | 41.2 | 33.3
  Strongly agree | 23.5 | 0

77. Secondary Outcome: Caregiver Questionnaire on Day 0 Post-treatment - Baby's Skin Looks Smooth in Areas Affected by Eczema
Description: Questions were answered after treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "In the areas affected by eczema, my baby's skin looks smooth".
Time Frame: 0 Days - Post-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 11.8 | 0
  Somewhat disagree | 41.2 | 66.7
  Neither agree nor disagree | 5.9 | 16.7
  Somewhat agree | 23.5 | 16.7
  Strongly agree | 17.6 | 0

78. Secondary Outcome: Caregiver Questionnaire on Day 0 Post-treatment - Baby's Skin Looks Healthy in Areas Affected by Eczema
Description: Questions were answered after treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "In the areas affected by eczema, my baby's skin looks healthy".
Time Frame: 0 Days - Post-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 5.9 | 0
  Somewhat disagree | 41.2 | 66.7
  Neither agree nor disagree | 17.6 | 16.7
  Somewhat agree | 23.5 | 16.7
  Strongly agree | 11.8 | 0

79. Secondary Outcome: Caregiver Questionnaire on Day 0 Post-treatment - Baby's Skin Feels Soft in Areas Affected by Eczema
Description: Questions were answered after treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "In the areas affected by eczema, my baby's skin feels soft".
Time Frame: 0 Days - Post-treatment
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 17 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 0 | 0
  Somewhat disagree | 29.4 | 50.0
  Neither agree nor disagree | 5.9 | 33.3
  Somewhat agree | 41.2 | 16.7
  Strongly agree | 23.5 | 0

80. Secondary Outcome: Caregiver Questionnaire on Day 3 - Skin Looks Smooth Overall
Description: Questions were answered after three days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Overall, my baby's skin looks smooth".
Time Frame: 3 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 0 | 0
  Somewhat disagree | 18.8 | 50.0
  Neither agree nor disagree | 12.5 | 0
  Somewhat agree | 50.0 | 50.0
  Strongly agree | 18.8 | 0

81. Secondary Outcome: Caregiver Questionnaire on Day 3 - Skin Looks Healthy Overall
Description: Questions were answered after three days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Overall, my baby's skin looks healthy".
Time Frame: 3 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 0 | 0
  Somewhat disagree | 6.3 | 16.7
  Neither agree nor disagree | 0 | 16.7
  Somewhat agree | 87.5 | 66.7
  Strongly agree | 6.3 | 0

82. Secondary Outcome: Caregiver Questionnaire on Day 3 - Skin Feels Soft Overall
Description: Questions were answered after three days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Overall, my baby's skin feels soft".
Time Frame: 3 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 0 | 0
  Somewhat disagree | 0 | 16.7
  Neither agree nor disagree | 18.8 | 16.7
  Somewhat agree | 56.3 | 50.0
  Strongly agree | 25.0 | 16.7

83. Secondary Outcome: Caregiver Questionnaire on Day 3 - Baby's Skin Looks Smooth in Areas Affected by Eczema
Description: Questions were answered after three days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "In the areas affected by eczema, my baby's skin looks smooth".
Time Frame: 3 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 0 | 16.7
  Somewhat disagree | 6.3 | 33.3
  Neither agree nor disagree | 12.5 | 0
  Somewhat agree | 75.0 | 50.0
  Strongly agree | 6.3 | 0

84. Secondary Outcome: Caregiver Questionnaire on Day 3 - Baby's Skin Looks Healthy in Areas Affected by Eczema
Description: Questions were answered after three days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "In the areas affected by eczema, my baby's skin looks healthy".
Time Frame: 3 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 0 | 16.7
  Somewhat disagree | 6.3 | 16.7
  Neither agree nor disagree | 6.3 | 33.3
  Somewhat agree | 75.0 | 33.3
  Strongly agree | 12.5 | 0

85. Secondary Outcome: Caregiver Questionnaire on Day 3 - Baby's Skin Feels Soft in Areas Affected by Eczema
Description: Questions were answered after three days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "In the areas affected by eczema, my baby's skin feels soft".
Time Frame: 3 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 0 | 16.7
  Somewhat disagree | 0 | 33.3
  Neither agree nor disagree | 12.5 | 16.7
  Somewhat agree | 68.8 | 33.3
  Strongly agree | 18.8 | 0

86. Secondary Outcome: Caregiver Questionnaire on Day 7 - Skin Looks Smooth Overall
Description: Questions were answered after seven days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Overall, my baby's skin looks smooth".
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 0 | 0
  Somewhat disagree | 6.3 | 16.7
  Neither agree nor disagree | 0 | 16.7
  Somewhat agree | 56.3 | 16.7
  Strongly agree | 37.5 | 50.0

87. Secondary Outcome: Caregiver Questionnaire on Day 7 - Skin Looks Healthy Overall
Description: Questions were answered after seven days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Overall, my baby's skin looks healthy".
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 6.3 | 0
  Somewhat disagree | 6.3 | 33.3
  Neither agree nor disagree | 0 | 0
  Somewhat agree | 50.0 | 16.7
  Strongly agree | 37.5 | 50.0

88. Secondary Outcome: Caregiver Questionnaire on Day 7 - Skin Feels Soft Overall
Description: Questions were answered after seven days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Overall, my baby's skin feels soft".
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 0 | 0
  Somewhat disagree | 0 | 0
  Neither agree nor disagree | 12.5 | 33.3
  Somewhat agree | 43.8 | 0
  Strongly agree | 43.8 | 66.7

89. Secondary Outcome: Caregiver Questionnaire on Day 7 - Baby's Skin Looks Smooth in Areas Affected by Eczema
Description: Questions were answered after seven days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "In the areas affected by eczema, my baby's skin looks smooth".
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 0 | 16.7
  Somewhat disagree | 6.3 | 33.3
  Neither agree nor disagree | 6.3 | 0
  Somewhat agree | 68.8 | 0
  Strongly agree | 18.8 | 50.0

90. Secondary Outcome: Caregiver Questionnaire on Day 7 - Baby's Skin Looks Healthy in Areas Affected by Eczema
Description: Questions were answered after seven days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "In the areas affected by eczema, my baby's skin looks healthy".
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 0 | 16.7
  Somewhat disagree | 6.3 | 33.3
  Neither agree nor disagree | 0 | 0
  Somewhat agree | 62.5 | 16.7
  Strongly agree | 31.3 | 33.3

91. Secondary Outcome: Caregiver Questionnaire on Day 7 - Baby's Skin Feels Soft in Areas Affected by Eczema
Description: Questions were answered after seven days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "In the areas affected by eczema, my baby's skin feels soft".
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 0 | 0
  Somewhat disagree | 0 | 50.0
  Neither agree nor disagree | 12.5 | 0
  Somewhat agree | 62.5 | 0
  Strongly agree | 25.0 | 50.0

92. Secondary Outcome: Caregiver Questionnaire on Day 7 - Child's Mood Over Past Week
Description: Questions were answered after seven days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Over this past week, what has your child's mood been?"
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Very happy | 37.5 | 33.3
  Somewhat happy | 37.5 | 16.7
  No change | 25.0 | 50.0
  Somewhat fussy | 0 | 0
  Very fussy | 0 | 0

93. Secondary Outcome: Caregiver Questionnaire on Day 7 - Child's Mood Upon Waking in Morning
Description: Questions were answered after seven days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Typically, how would you rate your child's mood when he/she wakes up in the morning?"
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Very happy | 25.0 | 0
  Somewhat happy | 50.0 | 16.7
  No change | 12.5 | 66.7
  Somewhat fussy | 12.5 | 16.7
  Very fussy | 0 | 0

94. Secondary Outcome: Caregiver Questionnaire on Day 7 - Child Wanted to Play Over Past Week
Description: Questions were answered after seven days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Over this past week, how much has your child wanted to play?"
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Less than last week | 0 | 0
  No difference | 56.3 | 50.0
  A little more | 18.8 | 16.7
  A lot more | 12.5 | 16.7
  All the time | 12.5 | 16.7

95. Secondary Outcome: Caregiver Questionnaire on Day 7 - Amount of Sleep Caregiver Got Over Past Week
Description: Questions were answered after seven days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Over this past week, how much sleep did you get at night?"
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
hours | 7.89 (1.626) | 7.42 (2.154)

96. Secondary Outcome: Caregiver Questionnaire on Day 7 - Number of Times Caregiver Woke Up
Description: Questions were answered after seven days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "How many times did you wake up during the night?"
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
number of times | 1.1 (0.89) | 1.7 (1.63)

97. Secondary Outcome: Caregiver Questionnaire on Day 7 - Amount of Time Caregiver Awake
Description: Questions were answered after seven days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "If you did wake up during the night, how much time were you awake (on average) before falling back asleep?"
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
hours | 0.32 (0.298) | 0.74 (0.754)

98. Secondary Outcome: Caregiver Questionnaire on Day 7 - Caregiver Energy Levels Over Past Week
Description: Questions were answered after seven days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Over this past week, how much energy have you had to engage with your family?"
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Less than last week | 0 | 0
  No difference | 37.5 | 66.7
  A little more | 37.5 | 16.7
  A lot more | 18.8 | 16.7
  All the time | 6.3 | 0

99. Secondary Outcome: Caregiver Questionnaire on Day 7 - How Rested Caregiver Felt Over Past Week
Description: Questions were answered after seven days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Over this past week, how rested have you felt?"
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Less than last week | 6.3 | 16.7
  No difference | 31.3 | 50.0
  A little more | 43.8 | 16.7
  A lot more | 12.5 | 16.7
  All the time | 6.3 | 0

100. Secondary Outcome: Caregiver Questionnaire on Day 7 - How Alert Caregiver Felt Over Past Week
Description: Questions were answered after seven days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Over this past week, how alert have you felt?"
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  I don't have an opinion | 0 | 0
  Less than last week | 0 | 0
  No difference | 50.0 | 66.7
  A little more | 37.5 | 16.7
  A lot more | 6.3 | 16.7
  All the time | 6.3 | 0

101. Secondary Outcome: Caregiver Questionnaire on Day 7 - How Productive Caregiver Felt Over Past Week
Description: Questions were answered after seven days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Over this past week, how productive have you been at work?"
Time Frame: 7 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 6
percentage of participants
  I don't have an opinion | 12.5 | 0
  Less than last week | 0 | 0
  No difference | 43.8 | 66.7
  A little more | 31.3 | 16.7
  A lot more | 6.3 | 16.7
  All the time | 6.3 | 0

102. Secondary Outcome: Caregiver Questionnaire on Day 14 - Skin Looks Smooth Overall
Description: Questions were answered after 14 days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Overall, my baby's skin looks smooth".
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 0 | 0
  Somewhat disagree | 0 | 20.0
  Neither agree nor disagree | 6.3 | 0
  Somewhat agree | 62.5 | 20.0
  Strongly agree | 31.3 | 60.0

103. Secondary Outcome: Caregiver Questionnaire on Day 14 - Skin Looks Healthy Overall
Description: Questions were answered after 14 days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Overall, my baby's skin looks healthy".
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 0 | 0
  Somewhat disagree | 0 | 20.0
  Neither agree nor disagree | 0 | 0
  Somewhat agree | 68.8 | 40.0
  Strongly agree | 31.3 | 40.0

104. Secondary Outcome: Caregiver Questionnaire on Day 14 - Skin Feels Soft Overall
Description: Questions were answered after 14 days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Overall, my baby's skin feels soft".
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 0 | 0
  Somewhat disagree | 0 | 0
  Neither agree nor disagree | 6.3 | 20.0
  Somewhat agree | 31.3 | 20.0
  Strongly agree | 62.5 | 60.0

105. Secondary Outcome: Caregiver Questionnaire on Day 14 - Baby's Skin Looks Smooth in Areas Affected by Eczema
Description: Questions were answered after 14 days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "In the areas affected by eczema, my baby's skin looks smooth".
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 0 | 0
  Somewhat disagree | 6.3 | 20.0
  Neither agree nor disagree | 0 | 20.0
  Somewhat agree | 62.5 | 20.0
  Strongly agree | 31.3 | 40.0

106. Secondary Outcome: Caregiver Questionnaire on Day 14 - Baby's Skin Looks Healthy in Areas Affected by Eczema
Description: Questions were answered after 14 days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "In the areas affected by eczema, my baby's skin looks healthy".
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 0 | 0
  Somewhat disagree | 0 | 20.0
  Neither agree nor disagree | 6.3 | 20.0
  Somewhat agree | 56.3 | 20.0
  Strongly agree | 37.5 | 40.0

107. Secondary Outcome: Caregiver Questionnaire on Day 14 - Baby's Skin Feels Soft in Areas Affected by Eczema
Description: Questions were answered after 14 days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "In the areas affected by eczema, my baby's skin feels soft".
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 6.3 | 0
  Somewhat disagree | 0 | 20.0
  Neither agree nor disagree | 6.3 | 20.0
  Somewhat agree | 37.5 | 0
  Strongly agree | 50.0 | 60.0

108. Secondary Outcome: Caregiver Questionnaire on Day 14 - Child's Mood Over Past Week
Description: Questions were answered after 14 days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Over this past week, what has your child's mood been?"
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
percentage of participants
  I don't have an opinion | 0 | 0
  Very happy | 12.5 | 20.0
  Somewhat happy | 25.0 | 40.0
  No change | 56.3 | 40.0
  Somewhat fussy | 6.3 | 0
  Very fussy | 0 | 0

109. Secondary Outcome: Caregiver Questionnaire on Day 14 - Child's Mood Upon Waking in Morning
Description: Questions were answered after 14 days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Typically, how would you rate your child's mood when he/she wakes up in the morning?"
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
percentage of participants
  I don't have an opinion | 0 | 0
  Very happy | 18.8 | 0
  Somewhat happy | 37.5 | 40.0
  No change | 31.3 | 40.0
  Somewhat fussy | 6.3 | 20.0
  Very fussy | 6.3 | 0

110. Secondary Outcome: Caregiver Questionnaire on Day 14 - Child Wanted to Play Over Past Week
Description: Questions were answered after 14 days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Over this past week, how much has your child wanted to play?"
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
percentage of participants
  I don't have an opinion | 0 | 0
  Less than last week | 0 | 0
  No difference | 43.8 | 40.0
  A little more | 18.8 | 0
  A lot more | 18.8 | 20.0
  All the time | 18.8 | 40.0

111. Secondary Outcome: Caregiver Questionnaire on Day 14 - Amount of Sleep Caregiver Got Over Past Week
Description: Questions were answered after 14 days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Over this past week, how much sleep did you get at night?"
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
hours | 7.99 (1.543) | 7.40 (1.710)

112. Secondary Outcome: Caregiver Questionnaire on Day 14 - Number of Times Caregiver Woke Up
Description: Questions were answered after 14 days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "How many times did you wake up during the night?"
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: number of times
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 15 | 5
number of times | 1.0 (1.07) | 1.6 (1.14)

113. Secondary Outcome: Caregiver Questionnaire on Day 14 - Amount of Time Caregiver Awake
Description: Questions were answered after 14 days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "If you did wake up during the night, how much time were you awake (on average) before falling back asleep?"
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
hours | 0.22 (0.385) | 0.87 (1.048)

114. Secondary Outcome: Caregiver Questionnaire on Day 14 - Caregiver Energy Levels Over Past Week
Description: Questions were answered after 14 days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Over this past week, how much energy have you had to engage with your family?"
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
percentage of participants
  I don't have an opinion | 0 | 0
  Less than last week | 0 | 0
  No difference | 43.8 | 60.0
  A little more | 31.3 | 0
  A lot more | 12.5 | 20.0
  All the time | 12.5 | 20.0

115. Secondary Outcome: Caregiver Questionnaire on Day 14 - How Rested Caregiver Felt Over Past Week
Description: Questions were answered after 14 days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Over this past week, how rested have you felt?"
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 15 | 5
percentage of participants
  I don't have an opinion | 0 | 0
  Less than last week | 0 | 0
  No difference | 40.0 | 60.0
  A little more | 40.0 | 20.0
  A lot more | 13.3 | 0
  All the time | 6.7 | 20.0

116. Secondary Outcome: Caregiver Questionnaire on Day 14 - How Alert Caregiver Felt Over Past Week
Description: Questions were answered after 14 days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Over this past week, how alert have you felt?"
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
percentage of participants
  I don't have an opinion | 0 | 0
  Less than last week | 0 | 0
  No difference | 50.0 | 60.0
  A little more | 37.5 | 20.0
  A lot more | 6.3 | 20.0
  All the time | 6.3 | 0

117. Secondary Outcome: Caregiver Questionnaire on Day 14 - How Productive Caregiver Felt Over Past Week
Description: Questions were answered after 14 days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "Over this past week, how productive have you been at work?"
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
percentage of participants
  I don't have an opinion | 6.3 | 0
  Less than last week | 0 | 0
  No difference | 50.0 | 60.0
  A little more | 31.3 | 0
  A lot more | 6.3 | 40.0
  All the time | 6.3 | 0

118. Secondary Outcome: Caregiver Questionnaire on Day 14 - Recommend Product
Description: Questions were answered after 14 days of treatment by participant's caregiver. Questions included overall look (smooth, healthy) and feel (soft, smooth) of participant's skin, and affected area's look (smooth, healthy) and feel (soft, smooth). The question is "I would recommend this product to another parent".
Time Frame: 14 Days
Population: The analysis was based on the intent-to-treat subjects who had data available at the specified time point.
Measure: Number; unit: percentage of participants
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Number analyzed (Participants) | 16 | 5
percentage of participants
  I don't have an opinion | 0 | 0
  Strongly disagree | 0 | 0
  Somewhat disagree | 0 | 20.0
  Neither agree nor disagree | 0 | 0
  Somewhat agree | 43.8 | 0
  Strongly agree | 56.3 | 80.0

ADVERSE EVENTS:
Time Frame: 14 ± 2 days, +30 days for serious adverse events.
Description: Adverse events were systematically collected beginning with the signing of the informed consent form and continuing at each study visit through Visit 7 (14 ± 2 days). Serious adverse events were reported through 30 days after product use. Spontaneously reported adverse events collected outside of the regularly scheduled visits were also recorded.
Arm/Group | 1% Colloidal Oatmeal Balm | EpiCeram Skin Barrier Emulsion
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/6
Other Adverse Events (participants affected / at risk) | 7/17 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1% Colloidal Oatmeal Balm (N=17) | EpiCeram Skin Barrier Emulsion (N=6)
Motion Sickness (Ear and labyrinth disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Frequent Bowel Movements (Gastrointestinal disorders) | 1 | 0
Teething (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 1
Ear Infection (Infections and infestations) | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 2 | 0
Scratch (Injury, poisoning and procedural complications) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 1 | 0
Keratosis Pilaris (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
A decision was made by the sponsor to terminate the study prior to enrolling 50 subjects as enrollment was not completed prior to the summer months, and the incidence of atopic dermatitis is low in the summer months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigators agreed not to publish the study results without prior sponsor approval.